CLINICAL TRIAL: NCT03920436
Title: Effects of Oral Ingestion of Drinking Water Using a Tumbler That Emits Far Infrared Rays at Room Temperature on Metabolic Profile in Adults: a RCT
Brief Title: Effects of Oral Ingestion of Drinking Water Using a Tumbler That Emits Far Infrared Rays on Metabolic Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor of Family Medicine, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-2018-035
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Problems

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrared water group (Experimental): This group takes drinking water using a tumbler that emits far infrared rays at room temperature for 8 weeks.
  Interventions: Dietary Supplement: infrared water group
- sham group (Sham Comparator): This group takes drinking water using a tumbler at room temperature for 8 weeks.
  Interventions: Dietary Supplement: sham group

INTERVENTIONS:
Dietary Supplement: infrared water group — This group takes 1,8 L of drinking water using a tumbler that emits far infrared rays at room temperature.
  Arms: Infrared water group
Dietary Supplement: sham group — This group takes 1,8 L of drinking water using a tumbler at room temperature.
  Arms: sham group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of oral ingestion of drinking water using a tumbler that emits far infrared rays at room temperature on metabolic profile in adults for 8 weeks.

DETAILED DESCRIPTION:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of oral ingestion of drinking water using a tumbler that emits far infrared rays at room temperature on metabolic profile in adults for 8 weeks; the safety of the compound are also evaluate. The Investigators examine lipid profile, glucose, liver and renal function at baseline, as well as after 4, 8 weeks of intervention. Thirty adults were administered either 1.8 L of drinking water using a tumbler that emits far infrared rays at room temperature or drinking water using a sham-tumbler each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older

Exclusion Criteria:

* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than twice the highest reference value
* serum creatinine ≥ 1.5 mg/dL)
* uncontrolled diabetes mellitus (a fasting glucose of >160 mg/dL)
* uncontrolled hypertension (BP > 160/100 mmHg)
* severe gastrointestinal symptoms
* alcohol abuser
* pregnant or lactating women
* allergic to the ingredient involved
* cardiocebrovascular diseases or any cancer during the six months prior to study
* smoker

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) | Change from baseline level of LDL-C at 8 weeks
  Change of LDL-C during 8 weeks

SECONDARY OUTCOMES:
aspartate transaminase (AST) | Change from baseline level of AST at 8 weeks
  Change of AST during 8 weeks
creatinine | Change from baseline level of creatinine at 8 weeks
  Change of creatinine during 8 weeks
homeostasis model assessment of insulin resistance (HOMA-IR) | Change from baseline level of HOMA-IR at 8 weeks
  Change of HOMA-IR during 8 weeks
body weight | Change from baseline level at 8 weeks
  Change of body weight during 8 weeks
free fatty acid | Change from baseline level at 8 weeks
  Change of free fatty acid during 8 weeks
alanine transaminase (ALT) | Change from baseline level of ALT at 8 weeks
  Change of ALT during 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea